CLINICAL TRIAL: NCT01705249
Title: Bleeding Profile With Continuous Hormone Replacement Therapy in Postmenopausal Women: A Prospective, Open, Multicenter Trial of Activelle® Treatment Following Switch From Trisekvens®
Brief Title: Bleeding Profile With Continuous Hormone Replacement Therapy of Activelle® in Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KLIM-1408
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Menopause; Healthy
MeSH Terms: interventions — Estradiol; Norethindrone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- estradiol / norethisterone acetate (Experimental)
  Interventions: Drug: 1.0 mg estradiol / 0.5 mg norethisterone acetate (NETA)

INTERVENTIONS:
Drug: 1.0 mg estradiol / 0.5 mg norethisterone acetate (NETA) — After a screening period of 12 weeks (three lunar months) in which the subjects still are on Trisekvens® followed by a treatment period of 24 weeks (six lunar months) in which the subjects are treated with Activelle®.

SUMMARY:
This study is conducted in Europe. The aim of this study is to investigate the bleeding profile after switch from Trisekvens® to Activelle® (1.0 mg estradiol / 0.5 mg norethisterone acetate (NETA)).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* At least 3 months on Trisekvens® before screening period
* Ability to understand and comply with the protocol requirements

Exclusion Criteria:

* Less than 12 months or more than 36 months postmenopausal judged by the Investigator
* Known, suspected, or past history of hormone dependent tumor/cancers
* Deep venous thrombosis, active thrombophlebitis, thromboembolic disorders, cerebrovascular accidents or past history of these conditions
* Ischemic heart disease or myocardial infarction within 6 months prior to randomization

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2001-08-14 (Actual); Primary Completion 2003-06-06 (Actual); Study Completion 2003-06-06 (Actual)

PRIMARY OUTCOMES:
Postmenopausal women's acceptance of bleeding | After 24 weeks of treatment

SECONDARY OUTCOMES:
Bleeding profile in postmenopausal women | After 24 weeks of treatment
Acceptance of hot flushes and breast tenderness | After 24 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (14):
- Norway (5):
  - Novo Nordisk Investigational Site, Kristiansand
  - Novo Nordisk Investigational Site, Kristiansund
  - Novo Nordisk Investigational Site, Larvik
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Trondheim
- Sweden (9):
  - Novo Nordisk Investigational Site, Borås
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Kungsbacka
  - Novo Nordisk Investigational Site, Linköping
  - Novo Nordisk Investigational Site, Norrköping
  - Novo Nordisk Investigational Site, Sigtuna
  - Novo Nordisk Investigational Site, Södertälje
  - Novo Nordisk Investigational Site, Stockholm
  - Novo Nordisk Investigational Site, Uddevalla

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com